CLINICAL TRIAL: NCT04725305
Title: BiZact Tonsillectomy
Brief Title: BiZact Tonsillectomy in the Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ronald Vilela, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-44399
Record Dates: First submitted 2020-11-26; First posted 2021-01-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Tonsillectomy; Tonsillitis Chronic; Hemorrhage; Postoperative Pain; Postoperative Hemorrhage; Surgery--Complications; Otorhinolaryngologic Diseases
Keywords: tonsillectomy; Bizact
MeSH Terms: conditions — Hemorrhage; Pain, Postoperative; Postoperative Hemorrhage; Otorhinolaryngologic Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two groups of participants will receive different interventions. One arm will receive the standard of care ( electrocautery) and the other group will receive the BIZACT method of tonsillectomy. The group allocation will be carried out by stratified randomization.
Who Masked: Participant
Masking Description: The participant will not be aware of the arm that the participate will be placed in- i.e. whether the tonsillectomy was carried out by electrocautery or using the BiZact device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BiZact (Experimental): A bipolar electrosurgical device that employs radiofrequency(RF) energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger
  Interventions: Device: BiZact
- Standard of care (Active Comparator): In electrocautery tonsillectomy (or diathermy) electric current from a radiofrequency generator is passed through the tissue between two electrodes. The resulting high temperature (400º-600ºC) cuts the tissue and simultaneously seals the blood vessels
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Device: BiZact — It has been described as describes a bipolar device that continuously measures impedance of clamped tissue, adjusting energy levels in real time and automatically stopping energy delivery when a seal is established. Their literature suggests the device permanently seals vessels up to 3mm with less thermal damage, resulting in less intraoperative blood loss, more efficient procedures, and possibly less pain
  Arms: BiZact
Procedure: Standard of care — This method would involve removal of tonsils using electrocautery technique
  Arms: Standard of care

SUMMARY:
This study has been designed to evaluate how effective the Bizact tonsillectomy device is in reducing operating time and complications that occur after surgery. This device operates in a different way than the standard device that is used for most tonsillectomies. In 2019, a study was conducted in 186 children and adults using this device in tonsillectomies. Results showed lower blood loss and shortened time in surgery. However, the rate for bleeding as a complication after surgery was the same as other procedures that are used in tonsillectomy

DETAILED DESCRIPTION:
Tonsillectomy is the second most common pediatric surgical procedure, with more than 280,000 performed in children under the age of 15 in the United States in 2010. The most common indications for tonsillectomy in children include recurrent infections and obstructive sleep apnea. While tonsillectomy in the pediatric population is generally safe and well-tolerated, post-operative complications are not uncommon, with post-operative pain, respiratory compromise, and post-tonsillectomy hemorrhage being chief among them.

Post-operative pain has been described as the main morbidity associated with tonsillectomy and is often ineffectively controlled. Pain beyond the initial 24-hour post-operative period has been noted to be worse with the use of electrocautery when compared to cold-knife dissection and snare tonsillectomy, perhaps attributable to the high levels of heat (400 °C to 600 °C) applied directly to the tonsillar area. Yet electrocautery remains one of the most frequently utilized tools due to its hemostatic effects through vessel coagulation at the time of dissection. Still, a recent large meta-analysis reported the rates of primary post-tonsillectomy hemorrhage (bleeding within the first 24 hours) at 2.4% and secondary post-tonsillectomy hemorrhage (beyond 24 hours) at 2.6%, suggesting that bleeding after tonsillectomy remains a relatively common occurrence. The search for a methodology that improves post-operative pain without increasing the risk of post-operative hemorrhage remains an active area of research.

Coblation, which creates an ionized plasma layer by passing a bipolar radio-frequency current through a medium of saline, offers another approach. The saline irrigation results in much less heat when compared to monopolar cautery, measuring approximately 40°C to 70°C. Coblation can be used in both subcapsular and intracapsular fashion. Subcapsular tonsillectomy with coblation has demonstrated a minimal decrease in pain, and may result in slightly higher rates of post-operative hemorrhage.

It has been pointed out that bipolar cautery could result in lower thermal injury and reduced blood loss, however tonsillectomy using traditional bipolar forceps leads to longer operative times. One group found that the use of BiClamp, a bipolar vascular sealing device originally designed for thyroidectomy, provided decreased operative times and less intraoperative bleeding compared to electrocautery. They noted, however, instances of posterior pillar perforation, which they attributed to curvature of the device that was designed for thyroid surgery, making dissection of the superior pole more difficult. Medtronic has now developed a similar device designed for use in tonsillectomy with a curved jaw meant to follow the contour of the tonsillar bed. In its marketing material for the recently developed BiZact , Medtronic describes a bipolar device that continuously measures the impedance of clamped tissue, adjusting energy levels in real-time and automatically stopping energy delivery when a seal is established. Their literature suggests the device permanently seals vessels up to 3mm with less thermal damage, resulting in less intraoperative blood loss, more efficient procedures, and possibly less pain.

In a pilot study of 186 patients, intraoperative blood loss was shown to be <1ml of blood loss in 71 cases (38.2%) and between 1 and 10ml of blood loss in 81 cases (43.5%). Post-operative hemorrhage rate of 4.3% is similar to rates described by other studies. BiZact tonsillectomy allows for a shortened operative time with a median time of 5.1 minutes. Other studies have shown other techniques to have a time duration of 21.6 minutes (electrocautery), 20.20 minutes (coblator), and 16.14 minutes (microdebrider).

In off label use of the device at our institution, data from surgeons using the device showed that surgeons perceived a relative improvement in following compared to standard tonsillectomy:

1. Less perceived thermal heat transfer to surrounding soft tissues
2. Left perceived blood loss
3. Superior ease of obtaining timely hemostasis
4. Faster operative time

ELIGIBILITY:
Inclusion Criteria:

* Tonsil hypertrophy with sleep disordered breathing
* Recurrent tonsillitis or pharyngitis
* Tonsil asymmetry or neoplasm
* Tonsil stones
* Must be able to take ibuprofen

Exclusion Criteria:

* Bleeding disorders such as von Willebrand's disease or hemophilia
* Down's Syndrome or other craniofacial syndromes
* Revision tonsillectomy cases

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Emergency room visits | 2 months
  Emergency room visits following tonsillectomy commonly involve poorly controlled pain, dehydration, and post-tonsillectomy hemorrhage. The investigators will tabulate the number of ER visits related to post-operative factors by reviewing charts of tonsillectomy patients two months post-operatively.
Intra-operative blood loss | Duration of surgery
  Intra-operative blood loss will be recorded in milliliters for all patients undergoing tonsillectomy using the BiZact device. Additionally, each surgeon using the Bi-zact device will maintain records of intra-operative blood loss in milliliters for tonsillectomies utilizing standard electrocautery for tonsillectomy.

SECONDARY OUTCOMES:
Post-tonsillectomy hemorrhage | 2 months
  Post-tonsillectomy hemorrhage is a known complication of tonsillectomy. The investigators will tabulate the incidence of post-tonsillectomy hemorrhage by reviewing emergency room visits in the post-operative period and through follow-up questionnaires at the first post-operative clinic visit.
Pain level | 14 days
  Patients will be asked to maintain a pain diary. The investigators will ask the parent or caretaker to document the Wong-Baker FACES Pain Rating Scale twice a day for fourteen days.
Pain medication documentation | 5 days
  Post-operative pain protocol at Texas Children's Hospital includes scheduled weight-based doses of ibuprofen every 6 hours for 5 days, acetaminophen every 4-6 hours as needed, and a one-time dose of dexamethasone as needed to be given on post-operative day 3, 4, or 5 for breakthrough pain. Patients are also instructed to use ibuprofen as needed for pain after the first 5 days. Participants will be instructed to maintain accurate records of use of acetaminophen and dexamethasone use, and use of ibuprofen beyond 5 days post-operatively
Operating time | Duration of procedure
  Operative time in minutes will be recorded for all patients undergoing tonsillectomy using the BiZact device. Additionally, each surgeon using the BiZact device will maintain records of operative time using standard electrocautery for tonsillectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall MJ, Schwartzman A, Zhang J, Liu X. Ambulatory Surgery Data From Hospitals and Ambulatory Surgery Centers: United States, 2010. Natl Health Stat Report. 2017 Feb;(102):1-15. PMID 28256998
- [Background] Rosenfeld RM, Green RP. Tonsillectomy and adenoidectomy: changing trends. Ann Otol Rhinol Laryngol. 1990 Mar;99(3 Pt 1):187-91. PMID 2178542
- [Background] De Luca Canto G, Pacheco-Pereira C, Aydinoz S, Bhattacharjee R, Tan HL, Kheirandish-Gozal L, Flores-Mir C, Gozal D. Adenotonsillectomy Complications: A Meta-analysis. Pediatrics. 2015 Oct;136(4):702-18. doi: 10.1542/peds.2015-1283. Epub 2015 Sep 21. PMID 26391937
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257
- [Background] Nunez DA, Provan J, Crawford M. Postoperative tonsillectomy pain in pediatric patients: electrocautery (hot) vs cold dissection and snare tonsillectomy--a randomized trial. Arch Otolaryngol Head Neck Surg. 2000 Jul;126(7):837-41. doi: 10.1001/archotol.126.7.837. PMID 10888995
- [Background] Jones DT, Kenna MA, Guidi J, Huang L, Johnston PR, Licameli GR. Comparison of postoperative pain in pediatric patients undergoing coblation tonsillectomy versus cautery tonsillectomy. Otolaryngol Head Neck Surg. 2011 Jun;144(6):972-7. doi: 10.1177/0194599811400369. Epub 2011 Apr 4. PMID 21493315
- [Background] Heidemann CH, Wallen M, Aakesson M, Skov P, Kjeldsen AD, Godballe C. Post-tonsillectomy hemorrhage: assessment of risk factors with special attention to introduction of coblation technique. Eur Arch Otorhinolaryngol. 2009 Jul;266(7):1011-5. doi: 10.1007/s00405-008-0834-2. Epub 2008 Oct 25. PMID 18953553
- [Background] Lee SW, Jeon SS, Lee JD, Lee JY, Kim SC, Koh YW. A comparison of postoperative pain and complications in tonsillectomy using BiClamp forceps and electrocautery tonsillectomy. Otolaryngol Head Neck Surg. 2008 Aug;139(2):228-34. doi: 10.1016/j.otohns.2008.04.004. PMID 18656720
- [Background] Pizzuto MP, Brodsky L, Duffy L, Gendler J, Nauenberg E. A comparison of microbipolar cautery dissection to hot knife and cold knife cautery tonsillectomy. Int J Pediatr Otorhinolaryngol. 2000 May 30;52(3):239-46. doi: 10.1016/s0165-5876(00)00293-7. PMID 10841953
- [Background] Medtronic Brief: More efficient tonsillectomies. Boulder Colorado, 2017. Retrieved from http://www.medtronic.com/content/dam/covidien/library/us/en/product/vessel-sealing/bizact-tonsillectomy-device-product-information-kit.pdf, 9/23/18.
- [Background] Krishnan G, Stepan L, Du C, Padhye V, Bassiouni A, Dharmawardana N, Ooi EH, Krishnan S. Tonsillectomy using the BiZact: A pilot study in 186 children and adults. Clin Otolaryngol. 2019 May;44(3):392-396. doi: 10.1111/coa.13273. Epub 2019 Feb 4. No abstract available. PMID 30576062